CLINICAL TRIAL: NCT04073706
Title: A Phase III Randomised Clinical Trial Comparing Sentinel Node Biopsy With No Retroperitoneal Node Dissection in Apparent Early-Stage Endometrial Cancer
Brief Title: Sentinel Node Biopsy in Endometrial Cancer
Acronym: ENDO-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDO-3
Record Dates: First submitted 2019-08-26; First posted 2019-08-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer Stage I; Sentinel Lymph Node; Surgery
Keywords: uterine cancer; sentinel node biopsy
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TH BSO with SNB (Experimental): Total Laparoscopic/Robotic Hysterectomy, Bilateral Salpingo-Oophorectomy (TH BSO) with Sentinel Node Biopsy (SNB) using Indocyanine Green (ICG)+/- Methylene Blue Dye (+/- omentectomy in high risk cell types) Note: If participants (≤45 years of age), have Grade 1 endometrial adenocarcinoma (EAC) with myometrial invasion <50% (by MRI) and wish to retain their ovaries a BSO may be omitted.
  Interventions: Procedure: TH BSO with SNB Note: If participants (≤45yo), Grade 1 endometrial adenocarcinoma with myometrial invasion <50%, wish to retain their ovaries a BSO may be omitted
- TH BSO without retroperitoneal node dissection (Active Comparator): Total Laparoscopic/Robotic Hysterectomy, Bilateral Salpingo-Oophorectomy (TH BSO) without retroperitoneal node dissection (+/- omentectomy in high risk cell types) Note: If participants (≤45 years of age), have Grade 1 endometrial adenocarcinoma (EAC) with myometrial invasion <50% (by MRI) and wish to retain their ovaries a BSO may be omitted.
  Interventions: Procedure: TH BSO without retroperitoneal node dissection Note: If participants (≤45yo), Grade 1 endometrial adenocarcinoma with myometrial invasion <50%, wish to retain their ovaries a BSO may be omitted

INTERVENTIONS:
Procedure: TH BSO with SNB Note: If participants (≤45yo), Grade 1 endometrial adenocarcinoma with myometrial invasion <50%, wish to retain their ovaries a BSO may be omitted — Removal of uterus, tubes and ovaries with a sentinel node biopsy. A tracer dye (ICG) +/- Methylene Blue Dye is injected into the surroundings of the primary tumour, it is transported via local lymphatic channels towards the draining lymphatic basin, and the first node that the tracer reaches is called the "sentinel node". These one or two nodes are thought to be first involved with cancer spread.
  Arms: TH BSO with SNB
Procedure: TH BSO without retroperitoneal node dissection Note: If participants (≤45yo), Grade 1 endometrial adenocarcinoma with myometrial invasion <50%, wish to retain their ovaries a BSO may be omitted — Removal of uterus, tubes and ovaries without retroperitoneal node dissection
  Arms: TH BSO without retroperitoneal node dissection

SUMMARY:
Endometrial cancer (EC) is the most common gynaecological cancer. Current treatment of EC typically includes removal of the uterus and to determine the extent of the disease (removal of fallopian tubes, ovaries & if required a lymph node dissection (surgical staging)). While lymph node dissection may be valuable to guide the need for adjuvant treatment (chemo or radiotherapy) after surgery, it has been a topic of controversy for the last 30 years. In some patients it causes morbidity, specifically lymphoedema. This recently has been replaced with sentinel node biopsy (SNB). It requires an injection of a dye into the cervix with specific equipment & surgical dissection of the lymph node in which the dye first becomes visible. Despite this promising proposition & similar to a lymph node dissection, the value to patients, cost effectiveness & potential harms (e.g. lymphedema) of SNB compared to no-node dissection in EC has never been established. Aim: determine the value of SNB for patients, the healthcare system and exclude detriment to patients using a randomised approach 1:1. Stage 1 - 444 patients. Stage 2 additional 316 patients.

Primary Outcome Stage 1:

Proportion of participants returning to usual daily activities at 12 months from surgery using the EQ-5D which will determine when women in both groups can return to their usual activities.

Primary Outcome Stage 2:

Treatment non-inferiority as evaluated by disease-free survival status at 4.5 years post-surgery, as measured by the time interval between the date of randomisation and date of first recurrence. Confirmation of recurrent disease will be ascertained through clinical assessment, radiological work-up and/or histological results.

DETAILED DESCRIPTION:
Hypothesis: The primary hypothesis is that SNB will not cause detriment to patients (lymphoedema, morbidity, loss of quality of life) and not increase costs compared to patients without a retroperitoneal node dissection. The secondary hypothesis is that disease-free survival in patients without retroperitoneal node dissection is not inferior to those receiving SNB.

Aims: To determine the value of SNB for patients, the healthcare system and to exclude detriment to patients.

Objectives:

Primary Stage 1:

To determine the recovery of participants (defined as incidence of adverse events, lower limb lymphoedema and health-related QOL) and to the healthcare system (cost) of Sentinel Node Biopsy (SNB) for the surgical treatment of endometrial cancer.

Primary Stage 2:

Compare disease-free survival at 4.5 years for participants randomised to receive hysterectomy, bilateral salpingo-oophorectomy with SNB compared to participants randomised to hysterectomy, bilateral salpingo-oophorectomy without retroperitoneal node dissection.

Secondary:

* Compare patterns of recurrence and overall survival (OS) between the groups
* Determine the cost-effectiveness of SNB
* Compare Patient Reported Outcomes (PROMS) between the groups at 12 months from surgery
* Compare Health Related Quality of Life (HRQL) and Fear of Recurrence between the groups at 12 months from surgery
* Compare perioperative outcomes (duration of surgery, length of hospital stay, intraoperative blood loss, blood transfusion requirements) and the incidence of intra- and postoperative adverse events within 12 months from surgery between the groups
* Compare lower limb lymphoedema at 12 months after surgery
* Compare the need for postoperative (adjuvant) treatments between groups
* Determine the impact of body composition and frailty on survival, quality of life, lymphoedema, peri-, intra- and postoperative outcomes
* Compare follow-up strategies (clinical vs symptom checklist)
* Translational Research - Trans-ENDO 3 - biobanking strategy - Compare the Molecular profile at 12 months from surgery between the groups

ELIGIBILITY:
Inclusion Criteria:

1. Females, over 18 years, with histologically confirmed primary epithelial cancer of the endometrium of any cell type or uterine carcinosarcoma (mixed malignant mullerian tumour);
2. Clinically stage I disease (disease confined to body of uterus);
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
4. Signed written informed consent;
5. Participant must meet criteria for a laparoscopic or robotic surgical approach as determined by the treating physician (e.g. suitable for TH BSO, ability to tolerate Trendelenberg positioning)
6. All available clinical evidence (physical examination findings, or medical imaging such as CT, MRI or ultrasound) demonstrates no evidence of extrauterine disease
7. Myometrial Invasion on MRI of not more than 50%. (Only if participant is <45yo, has ONLY Grade 1 EAC and wishes to retain their ovaries).
8. Negative (serum or urine) pregnancy test ≤ 30 days of surgery in pre-menopausal women and women < 2 years after the onset of menopause.

Exclusion Criteria:

1. Evidence of extrauterine disease (apparent involvement of cervix, vagina, parametria, adnexa, lymph nodes, bladder, bowel or distant sites) by clinical examination and/or through medical imaging.
2. Enlarged retroperitoneal pelvic and/or aortic lymph nodes (>1 cm) on medical imaging;
3. Estimated life expectancy of less than 6 months;
4. Patients who have absolute contraindications for adjuvant radiotherapy and/or chemotherapy;
5. Patients who have previously received radiation treatment to the pelvis
6. Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator);
7. Patient compliance and geographic proximity that do not allow adequate follow-up;
8. Patients with allergy to Indocyanine Green (ICG)
9. Patients who have had previous retroperitoneal surgery
10. Patients who require a retroperitoneal (pelvic +/- para-aortic) lymph node dissection (lymphadenectomy)
11. Other prior malignancies <5 years before inclusion, except for successfully treated keratinocyte skin cancers, or ductal carcinoma of the breast insitu
12. Uterine perforation during endometrial tissue sampling

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Return to usual activities | 12 months from surgery
  Proportion of participants returning to usual daily activities at 12 months from surgery using the EQ-5D which will determine when women in both groups can return to their usual activities.
Stage 2: Disease Free Survival | 4.5 years from surgery
  Compare disease-free survival for participants randomised to receive hysterectomy, bilateral salpingo-oophorectomy with SNB compared to participants randomised to hysterectomy, bilateral salpingo-oophorectomy without retroperitoneal node dissection

SECONDARY OUTCOMES:
Cost Effectiveness using QALYs using EuroQoL-5D (EQ-5D) Questionnaire | 12 months from surgery
  An assessment will be performed on the cost-effectiveness of TH + SNB relative to TH alone, calculated as the incremental cost per unit of improvement in functional outcome, measured in terms of the primary outcome. This will assess how much more money the proposed intervention will cost the health system and society, and whether this represents a sound investment in terms of the improvement in quality of life. We will also measure the quality-adjusted life years (QALYs) gained with the intervention and use this to undertake a cost-utility analysis. The QALY calculations will be based on health status measures for trial participants, with valuations of changes in health status and quality of life based on the EQ-5D
Cost Effectiveness measuring Intervention costs | 12 months from surgery
  An assessment will be performed on the cost-effectiveness of TH + SNB relative to TH alone, calculated as the incremental cost per unit of improvement in functional outcome, measured in terms of the primary outcome. This will assess how much more money the proposed intervention will cost the health system and society.
Cost Effectiveness measuring GP and specialist consultations | 12 months from surgery
  An assessment will be performed on the cost-effectiveness of TH + SNB relative to TH alone, calculated as the incremental cost per unit of improvement in functional outcome, measured in terms of the primary outcome. This will assess how much more money the proposed intervention will cost the health system and society, and whether this represents a sound investment in terms of the improvement in quality of life.
Cost Effectiveness measuring radiology and imaging requirements | 12 months from surgery
  An assessment will be performed on the cost-effectiveness of TH + SNB relative to TH alone, calculated as the incremental cost per unit of improvement in functional outcome, measured in terms of the primary outcome. This will assess how much more money the proposed intervention will cost the health system and society.
Cost Effectiveness measuring prescriptions and over the counter medicine requirements | 12 months from surgery
  An assessment will be performed on the cost-effectiveness of TH + SNB relative to TH alone, calculated as the incremental cost per unit of improvement in functional outcome, measured in terms of the primary outcome. This will assess how much more money the proposed intervention will cost the health system and society, and whether this represents a sound investment in terms of the improvement in quality of life.
Cost Effectiveness measuring community and health service requirements and days off work and informal care required by family and friends using a combination of the Health Services Questionnaire and clinical files | 12 months from surgery
  An assessment will be performed on the cost-effectiveness of TH + SNB relative to TH alone, calculated as the incremental cost per unit of improvement in functional outcome, measured in terms of the primary outcome. This will assess how much more money the proposed intervention will cost the health system and society, and whether this represents a sound investment in terms of the improvement in quality of life.
Cost Effectiveness: direct costs using a bottom-up approach by recording the volume of resource use in both groups of the trial, and then applying a unit cost to each component | 12 months from surgery
  Direct costs wukk be ibtained for smaples of participants, stratified by hospital, operation and outcome to assess the cost-effectiveness of TH + SNB relative to TH alone, calculated as the incremental cost per unit of improvement in functional outcome, measured in terms of the primary outcome. This will assess how much more money the proposed intervention will cost the health system and society.
Perioperative Outcomes: Adverse Events | 12 months from surgery
  Compare perioperative outcomes and the incidence of intra- and postoperative adverse events within 12 months from surgery between groups using Common Terminology Criteria for Adverse Events (CTCAE version 5)
Perioperative Outcomes: Length of Surgery | At time of surgery
  Compare the length of surgery between the two groups. This will be recorded in hh:mm on the surgery form.
Perioperative Outcomes: Blood Loss during Surgery | At time of surgery
  Compare the blood loss between the two groups during surgery. This will be recorded in ml.
Perioperative Outcomes: Blood Transfusion Requirements during Surgery | At time of surgery
  Compare the blood transfusion requirements between the two groups. This will be recorded in units and recorded on the Surgery Form and the Concomitant Medication Form.
Perioperative Outcomes: Length of Hospital Stay | At time of discharge from hospital following surgery
  Compare the length of hospital stay between the two groups. The duration will be measured in days. Date of surgery being day 0.
Health Related Quality of Life and Fear of Recurrence | 12 months from surgery
  Change in Quality of Life using Functional Assessment of Cancer General (FACT-EN), Fear of Recurrence and PROMS between baseline and 1 year after surgery
Incidence of Lymphedema | 12 months from surgery
  Compare lower limb lymphedema between groups
Adjuvant Treatment Requirements | 12 months from surgery
  Compare the need for postoperative (adjuvant) treatments between groups and evaluate the impact of SNB on clinical decisions regarding adjuvant treatment. Any chemotherapy or radiation therapy required will be recorded on specific chemotherapy or radiation forms. Chemotherapy will be recorded in mg received and number of doses required including start/end dates. Radiation treatment received will be recorded as total dose of Gy and how many fractions, including start and end dates.
Value of Molecular Biomarkers | 24 months from surgery
  Translational Research - Compare Molecular profile from surgery between the groups that require adjuvant therapy for 24 months.
Value of Molecular Biomarkers | 12 months from surgery
  Translational Research - Compare the Molecular profile of Germline DNA at 12 months from surgery between the groups
Value of Molecular Biomarkers | 12 months from surgery
  Translational Research - Compare the Molecular profile of Circulating Tumour DNA at 12 months from surgery between the groups
Value of Molecular Biomarkers | 12 months from surgery
  Translational Research - Compare the Molecular profile of Plasma at 12 months from surgery between the groups
Value of Molecular Biomarkers | 12 months from surgery
  Translational Research - Compare the Molecular profile of Serum at 12 months from surgery between the groups
Overall Survival | 4.5 years from surgery
  Compare overall survival for participants randomised to receive hysterectomy, bilateral salpingo-oophorectomy with SNB compared to participants randomised to hysterectomy, bilateral salpingo-oophorectomy without retroperitoneal node dissection
Patterns of Recurrence - date and localization of 1st recurrence | 4.5 years from surgery
  Date and localization of 1st recurrence as confirmed histologically and/or radiologically - Compare these patterns of recurrences between the groups. These will also be adjudicated by an independent committee to ensure accuracy of documented recurrence
Impact of body composition (sarcopenia) on surgical complications, recovery and overall survival | 4.5 years from surgery
  Body mass measures are practical & sensitive for predicting health risks & outcomes. Sarcopenia is defined as loss of skeletal muscle mass & strength. It's been found to be associated with procedure-related morbidity, survival in cancer patients and increased use of healthcare. The concurrent appearance of low muscle mass with high adiposity (sarcopenic obesity) is common in people with chronic diseases. The trial will determine the role sarcopenia has on participants pre-operatively (via CT images & Bioimpedance Spectroscopy (BIS - if available at site) & postoperatively using the BIS in regard to survival in gynaecological malignancies, if it is a predictive factor for treatment adverse events & participants tolerability of treatment & compare diagnostic methods to determine medical fitness for surgery. BIS sends non-detectable electrical currents, at a range of frequencies through the body allowing precise measurement & analysis of impedance to currents by extracellular fluid
Impact of frailty on surgical complications, recovery and overall survival | 4.5 years from surgery
  It has been reported consistently that frailty has a significant impact on the occurrence of adverse postoperative outcomes. Therefore, measuring frailty is important to estimate risks, determine the best treatment options, and to aid diagnosis and care planning. Frailty will be measured prior to surgery suing the validated tool - Frailty Phenotype. This may determine the impact frailty has on survival, quality of life, lymphedema, peri-, intra- and postoperative outcomes
Follow-Up Strategies | 4.5 years from surgery
  Current institutional & clinical guidelines suggest patients need to be seen at regular follow up visits. The risk of developing a recurrence is higher within the initial period after surgery & the majority of recurrences develop within those first 3 years. Participants will ideally be seen 3 monthly for the first 3 years & 6 monthly until 4.5 years. The objective of follow up is that local recurrences from endometrial cancer are potentially curable. It helps to diagnose local recurrences as early as possible so that they are amenable for curative or effective palliative management. We will compare these clinical findings to a symptom checklist that will be completed by participants every 3 months from surgery until 4.5 years. This records patient reported symptoms that may indicate a recurrence. Comparing these findings should determine effective follow up strategies for this group of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, Prof, Study Chair — Director, Queensland Centre for Gynaecological Cancer Research
Locations (19):
- Houston Methodist Hospital, Houston, Texas, United States
- Hospital Britanico, Buenos Aires, Ciudad Autónoma de Buenos Aires (caba), Argentina
- Australia (11):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - The Wesley Hospital, Auchenflower, Queensland
  - Buderim Private Hospital, Buderim, Queensland
  - North West Private Hospital, Everton Park, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Hospital, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - St Andrews War Memorial Hospital, Spring Hill, Queensland
  - Mercy Hospital for Women, Heidelberg, Victoria
  - Royal Women's Hospital, Parkville, Victoria
- Brazil (3):
  - Hospital de Base, São José do Rio Preto, São Paulo
  - Fundacao Antonio Prudente, AC Camargo Cancer Center, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
- Centro de tratamiento e investigación sobre Cáncer Luis Carlos Sarmiento Angulo, Bogotá, Bogotá, Distrito Capital, Colombia
- Azienda Sanitaria Universitaria Friuli Centrale (ASUFC), Udine, Via Pozzuolo, Italy
- National University Hospital and National University Cancer Institute, Singapore, NUH Zone B, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Obermair A, Nicklin J, Gebski V, Hayes SC, Graves N, Mileshkin L, Lin MY, Beale P, Baxter E, Robledo K, Salomon C, Hanna GB, Janda M. A phase III randomized clinical trial comparing sentinel node biopsy with no retroperitoneal node dissection in apparent early-stage endometrial cancer - ENDO-3: ANZGOG trial 1911/2020. Int J Gynecol Cancer. 2021 Dec;31(12):1595-1601. doi: 10.1136/ijgc-2021-003029. Epub 2021 Nov 2. PMID 34728527